CLINICAL TRIAL: NCT06465017
Title: ImmunoPET Targeting Trophoblast Cell-Surface Antigen 2 (Trop-2) in Thyroid Cancer and Compared With 18F-FDG and 68Ga-FAPI
Brief Title: ImmunoPET Targeting Trophoblast Cell-Surface Antigen 2 (Trop-2) in Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XMYY-2024KY195
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-03

CONDITIONS: Tumor; Solid Tumor; Thyroid Cancer; Positron-Emission Tomography
Keywords: Tumor; Solid; Positron-Emission Tomography; Trop-2; Diagnosis
MeSH Terms: conditions — Neoplasms; Thyroid Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-THP-Trop2 VHH (Experimental): Each subject receives a single intravenous injection of 68Ga-THP-Trop2 VHH and undergoes PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: standard-of-care imaging (18F-FDG and 68Ga-FAPI PET/CT), 68Ga-THP-Trop2 VHH PET/CT

INTERVENTIONS:
Diagnostic Test: standard-of-care imaging (18F-FDG and 68Ga-FAPI PET/CT), 68Ga-THP-Trop2 VHH PET/CT — Each subject receives a single intravenous injection of standard-of-care imaging radiopharmaceuticals (18F-FDG and 68Ga-FAPI) and 68Ga-THP-Trop2 VHH, and undergoes PET/CT imaging within the specified time.

SUMMARY:
The objective of the study is to construct a noninvasive approach 68Ga-THP-Trop2 VHH PET/CT to detect the Trop-2 expression of tumor lesions in patients with thyroid cancer and to identify patients benefiting from Trop-2 targeting antibody-drug conjugate treatment.

DETAILED DESCRIPTION:
As a new trophoblast cell-surface antigen 2 (Trop-2) targeting PET radiotracer, 68Ga-THP-Trop2 VHH is promising as an excellent imaging agent applicable to various cancers. In this research, subjects with thyroid cancer or highly suspected recurrence detection underwent contemporaneous 68Ga-THP-Trop2 VHH and standard-of-care imaging (18F-FDG and 68Ga-FAPI PET/CT) either for an initial assessment or for metastases or highly suspected recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The numbers of positive tumor lesions of standard-of-care imaging and 68Ga-THP-Trop2 VHH PET/CT were recorded by visual interpretation. The diagnostic accuracy of 68Ga-THP-Trop2 VHH was calculated and compared to standard-of-care imaging.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or older);
* Patients with newly diagnosed, highly suspected recurrence or previously treated metastases of thyroid cancer (supporting evidence may include MRI, CT, tumor markers, and pathology report);
* Patients who had scheduled both standard-of-care imaging (18F-FDG and 68Ga-FAPI PET/CT) and 68Ga-THP-Trop2 VHH PET/CT scans;
* Patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* Patients with pregnancy;
* The inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Diagnostic efficacy | 2 years
  The sensitivity, specificity, and accuracy of standard-of-care imaging (18F-FDG and 68Ga-FAPI PET/CT) and 68Ga-THP-Trop2 VHH PET/CT were calculated and compared to evaluate the diagnostic accuracy.

SECONDARY OUTCOMES:
Number of lesions | 2 years
  The numbers of positive primary and metastatic lesions of standard-of-care imaging (18F-FDG and 68Ga-FAPI PET/CT) and 68Ga-THP-Trop2 VHH PET/CT were recorded by visual interpretation.
SUV | 2 years
  Standardized uptake value (SUV) of standard-of-care imaging (18F-FDG and 68Ga-FAPI PET/CT) and 68Ga-THP-Trop2 VHH PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China